CLINICAL TRIAL: NCT04687995
Title: The Tragal Perichondrium Versus the Pretragal Fascial Grafts for Endoscopic Myringoplasty: Comparative Study
Brief Title: Tragal Perichondrium Versus Pretragal Fascial (SMAS) Graft for Endoscopic Myringoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hazem Gamal Noreldein, Resident doctor in otolaryngology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endoscopic myringoplasty
Record Dates: First submitted 2020-09-26; First posted 2020-12-29 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tragal preichondrium graft (Active Comparator): Tragal perichodrium graft for endoscopic myringoplasty as a reference graft
  Interventions: Procedure: Endoscopic myringoplasty
- pretragal ( SMAS) fascia graft (Active Comparator): pretragal ( SMAS) fascia graft for endoscopic myringoplasty as a new graft
  Interventions: Procedure: Endoscopic myringoplasty

INTERVENTIONS:
Procedure: Endoscopic myringoplasty — Endoscopic myringoplasty by using two different grafts one each time

SUMMARY:
1. Examine the treatment outcomes of the pretragal (SMAS) fascia as a new graft when used in endoscopic myringoplasty.
2. Compare the results when using the tragal pericondrium as a graft in endoscopic myringoplasty regarding donor site and success.

DETAILED DESCRIPTION:
The exclusive transcanal endoscopic tympanoplasty technique emerged in the1990s : it provides a more direct and wider surgical viewing angle, largely reduces the necessity for a traumatic postauricular incision. Some otolgists have adopted this technique using the nearby tragal perichondrium/cartilage graft. The tragus has a pivotal function in reconstruction in ear surgery. The superficial musculoaponeurotic system (SMAS) was first introduced by Mits and Peyroniein1976. It is located in the mid-face overlying the parotid gland and mimic muscles, It connects the dermis and the muscles, acting as a unique motor unit to produce facial expressions. The SMAS graft has great potential because it is accessible from the least invasive transcanal route of tympanoplasty, and is located away from the vital structures.

ELIGIBILITY:
Inclusion Criteria:

1. Above 16 yrs old and less than 50 yrs old.
2. Clinically diagnosed central tympanic membrane perforations or chronic suppurative otitis media (tubo-tympanic).
3. Dry ear: no otorrhea without medication for at least 1 month.
4. Hearing loss gap not more than 50dB

Exclusion Criteria:

1. Age less than 16 or more than 50.
2. Discharging (active) central perforations.
3. Unsafe CSOM with cholesteatoma.
4. Suspected ossicular pathology in safe CSOM if the gap > 50dB.
5. Previous ear surgery.
6. Patients unfit for surgery or having chronic medical illness.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
comparison of tragal perichondrium versus pretragal fascial (SMAS) graft for endoscopic myringoplasty | Baseline
  comparison of results when using tragal perichondrium versus pretragal fascial (SMAS) graft for endoscopic myringoplasty success rate by audiological evaluation by using audiotympanogram

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin MY, Chang TS, Liao JB. The Pretragal Superficial Musculoaponeurotic System Fascia: A New Graft Material for Transcanal Tympanoplasty. Otol Neurotol. 2020 Jun;41(5):644-653. doi: 10.1097/MAO.0000000000002599. PMID 32080032